CLINICAL TRIAL: NCT04395209
Title: Muscle Strength Loss In Stroke Individuals - Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Suat EREL, prof. dr., Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pamukkale Uni
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Stroke Rehabilitation

STUDY DESIGN:
Intervention Model Description: individuals with stroke and healthy subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroke individuals (Experimental)
  Interventions: Other: assesment
- healthy individuals (Active Comparator)
  Interventions: Other: assesment

INTERVENTIONS:
Other: assesment — muscle strength assessment in stroke individuals

SUMMARY:
ABSTRACT The muscle strength (MS) is necessary to overcome the resistance encountered during the activity. The present study aims to determine MS loss in stroke individuals (SI). 33 SI and 33 healthy individuals (HI) were included in this study. MS and handgrip force were assessed using a power track dynamometer and Jamar hand dynamometer, respectively. The total MS of the HI was calculated by summing the muscle strength of the trunk, lower and upper extremities. In the SI, the muscle strength of the trunk, unaffected upper and lower extremities were summed to calculate the total MS. To compare MS of unaffected sides (US) between groups, 27 SI who was dominant and not affected on the right side and 33 HI who was dominant on the right side were used.

ELIGIBILITY:
Inclusion Criteria:

* for patient with stroke
* Between 30-65 ages
* Diagnosed with stroke chronic stroke patients (diagnosed with a stroke at least 6 months ago)

for healthy individuals

* 30-65 ages
* healthy individuals

Exclusion Criteria for patient with stroke

* patient with an additional neurological disease to stroke
* patients with orthopedic problems,
* patients with mental and communication impairments
* patients who scored more than 3 points for the Modified Rankin Scale for healthy individuals;
* who had active sporting life

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Loss In Stroke Individuals - Control Study | 24 week
  muscle strength of stroke individuals was assesed by power track hand held dynamometer and The Jamar Hand dynamometer, And recorded in newton.

CONTACTS AND LOCATIONS:
Locations (1):
- University Address, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No